CLINICAL TRIAL: NCT01584076
Title: Recovery From Amblyopia With Cholinesterase Inhibitors
Brief Title: Treatment of Residual Amblyopia With Donepezil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Carolyn Wu, Assistant Professor of Ophthalmology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00002887
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Amblyopia
Keywords: Amblyopia; Donepezil
MeSH Terms: conditions — Amblyopia | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donepezil (Experimental)
  Interventions: Drug: Donepezil; Other: Patching

INTERVENTIONS:
Drug: Donepezil — Oral Donepezil Daily
  Initial Dosage: Donepezil 5 mg tablets will be used. 1/2 tablet (≈2.5 mg)/day for 8 to 17 year olds OR 1 tablet (5 mg)/day for ≥18 year olds.
  Dosage Escalation: Donepezil may be increased by 1/2 tablet (≈2.5 mg)/day every 4 weeks if the amblyopic eye visual acuity has not improved by ≥5 letters or 1 logMAR line to a maximum dosage of 1 1/2 tablets (≈7.5 mg)/day for 8 to 17 year olds OR 2 tablets (10 mg)/day for ≥18 year olds.
  Other Names: Aricept
Other: Patching — Patching: 2 hours of daily patching will also be prescribed for 8 to 17 year olds only.

SUMMARY:
Amblyopia is the leading cause of monocular visual impairment in children and adults. Despite conventional treatment with patching or eye drops, many older children and adults do not achieve normal vision in the amblyopic eye.

Donepezil is an acetylcholinesterase inhibitor that increases levels of the neurotransmitter acetylcholine in the brain. Use of acetylcholinesterase inhibitors has been demonstrated by the Hensch lab (Department of Neurology, FM Kirby Neurobiology Center) at Boston Children's Hospital to improve vision and reverse amblyopia in animal models.

The purpose of this study is to evaluate the efficacy of oral donepezil as treatment for residual amblyopia (20/50 - 20/400) in patients 8 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥8 years
2. Amblyopia associated with strabismus and/or anisometropia
3. Amblyopic eye visual acuity of 20/50 - 20/400
4. Sound eye visual acuity of ≥20/25
5. For 8 to 17 year olds, current amblyopia treatment of at least 2 hours of daily patching for at least 4 weeks during the pre-enrollment period with no improvement in best-corrected amblyopic eye visual acuity (<5 letters or 1 logMAR line between 2 consecutive visual acuity measurements at least 4 weeks apart while on current treatment)
6. For ≥18 year olds, history of prior amblyopia treatment with patching
7. Wearing optimal optical correction with stable amblyopic eye visual acuity (<5 letters or 1 logMAR line of improvement during 2 consecutive visual acuity measurements at least 4 weeks apart)
8. Complete eye examination within 6 months prior to enrollment
9. Available for at least 6 months of follow-up, have access to a phone, and willing to be contacted by clinical staff
10. Likely to comply with prescribed treatment and unlikely, if applicable, to continue to improve with 2 hours of daily patching alone

Exclusion Criteria:

1. Myopia more than -6.00 D spherical equivalent
2. Presence of associated findings that could cause reduced visual acuity
3. Previous intraocular or refractive surgery
4. Strabismus surgery planned within 22 weeks
5. Current vision therapy or orthoptics
6. Treatment with topical atropine within the past 4 weeks
7. Presence of cardiac condition, asthma, obstructive pulmonary disease, seizure disorder, urinary incontinence, and/or peptic ulcer disease receiving concurrent NSAIDs
8. History of gastrointestinal bleeding from peptic ulcer disease
9. Known psychological problems
10. Known skin reaction to patch or bandage adhesives for 8 to 17 year olds
11. Known allergies or contraindications to the use of acetylcholinesterase inhibitors
12. Prior acetylcholinesterase inhibitor treatment
13. Current use of medication for the treatment of ADHD or psychological disorders
14. Inability to swallow pills equivalent in size to the 5 mg donepezil tablet
15. Females who are pregnant, lactating, or intending to become pregnant within the next 6 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Amblyopia Eye Visual Acuity Improvement | 22 weeks after enrollment
  Study treatment will last for 12 weeks. Primary outcome measure is analysis of the proportion of subjects with improvement in amblyopic eye visual acuity of ≥ 15 letters or 3 logMAR lines at 22 weeks after 10 weeks off study treatment.

SECONDARY OUTCOMES:
Amblyopic Eye Visual Acuity | 4, 8, 12, and 22 weeks after enrollment
  Analysis of amblyopia eye visual acuity measured at each visit.
Recurrence of Amblyopia after 10 Weeks Off Study Treatment | 22 weeks after enrollment
  Study treatment will be discontinued after 12 weeks. Amblyopic eye visual acuity at 12 weeks and 22 weeks will be compared. Analysis of the proportion of subjects with recurrence of amblyopia after 10 weeks off study treatment.
Adverse Events | 4, 8, 12, and 22 weeks after enrollment
  Analysis of the proportion of subjects reporting adverse events.
Adverse Events Requiring Discontinuation of Study Treatment | 4, 8, and 12 weeks after enrollment
  Analysis of the proportion of subjects requiring discontinuation of study treatment secondary to adverse events.
Completion of Study Treatment | 12 weeks after enrollment
  Analysis of the proportion of subjects completing study treatment.
Sound Eye Visual Acuity | 22 weeks after enrollment
  Analysis of sound eye visual acuity at 22 weeks to assess any adverse effect on the occluded eye.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Wu, MD, Principal Investigator — Boston Children's Hospital; David G. Hunter, MD, PhD, Principal Investigator — Boston Children's Hospital; Bharti Gangwani, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Children's Hospital at Waltham, Waltham, Massachusetts
  - Boston Children's Physicians South, Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morishita H, Miwa JM, Heintz N, Hensch TK. Lynx1, a cholinergic brake, limits plasticity in adult visual cortex. Science. 2010 Nov 26;330(6008):1238-40. doi: 10.1126/science.1195320. Epub 2010 Nov 11. PMID 21071629